CLINICAL TRIAL: NCT00367263
Title: A Randomized Cross-Over Design Study Evaluating a Traditional Paper Symptom Diary vs. the VOCEL Mobile Diary in Subjects 12 Years and Older With Mild to Moderate Persistent Asthma Receiving Ciclesonide MDI (Alvesco) 80 ug BID
Brief Title: Evaluation of Traditional Paper Symptom Diary vs. the VOCEL Mobile Diary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergy & Asthma Medical Group & Research Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICLE-L-01335
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2007-05-02 (Estimated); Status verified 2007-04

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alvesco (Ciclesonide) 160 ug/day

SUMMARY:
This study is designed to evaluate a traditional paper symptom diary system versus the VOCEL Mobile Diary. Subjects will be issued in a random order each system and asked their preference at the end of their participation.

DETAILED DESCRIPTION:
Inflammation is the underlying pathophysiologic process causing asthma. Inhaled corticosteroids are the first drugs of choice for treatment. Monotherapy with an ICS is most often sufficient and, along with an as needed short acting bronchodilator agent, the most cost effective method for managing patients with mild-moderate persistent asthma.

Alvesco, the ICS ciclesonide delivered in a solution via a HFA metered dose inhaler, has been shown to be effective and safe for the treatment of persistent asthma. This study will attempt to further document these attributes in patients with mild-moderate persistent asthma.

The collection of patient reported data can be accomplished in a number of ways. The standard system in asthma trials is daily diaries transcribed on paper forms. While useful in many studies, this system lacks the ability to remind subject of reporting time, to time stamp when the report is done and note at the time of report completion to the subject, areas that are incomplete, and to remind patients when to take their study medication. Because of these inadequacies, newer electronic data collection systems are being developed. One of these, the VOCEL Mobile Diary system, will be compared with the standard paper reporting method for abilities to document efficacy, safety, compliance and convenience.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 12 years of age and older. Females will be eligible only if they are:

   1. Surgically sterilized, post-menopausal (>1 year), abstinent, or practicing adequate method of birth control, and if they have a
   2. Negative urine pregnancy test (females of childbearing potential)
2. History of mild to moderate persistent asthma for at least 6 months as defined by NIH NHLBI April 19971.

At Visit 1 (Screening) treatment of subjects for the lat 30 days prior to screening must be:

1. No inhaled corticosteroid therapy. Previous use of leukotriene receptor antagonists, and/or cromones, in addition to short acting bronchodilators are allowed.) Or,
2. Inhaled corticosteroid therapy in monotherapy or in combination with a long acting beta agonist (LABA).

Exclusion Criteria:

1. Female subjects who are pregnant or trying to become pregnant
2. Breast feeding
3. Viral or bacterial respiratory tract infection within the last 14 days
4. Tobacco smoking within the previous 6 months or greater than a lifetime 10 pack-year smoking history
5. History of glaucoma, cataracts (lens opacities), retinal disease, or blindness
6. Any serious concomitant disease such as cancer or serious renal, hepatic, cardiac, immunodeficiency, neurological, psychiatric, or other disease
7. Any medical condition that, in the judgment of the investigator, might interfere with the study, require treatment or make implementation of the protocol or interpretation of the study results difficult
8. Active or quiescent tuberculosis infections of the respiratory tract
9. History of chronic bronchitis, COPD or emphysema
10. History of alcohol abuse (more than 2 drinks/day on average) or drug abuse within the past 2 years
11. Treatment with any investigational drug within the past 30 days
12. Subjects can be on maintenance immunotherapy but cannot have begun an immunotherapy regimen or have had a change in their immunotherapy regimen within 30 days prior to screening (Visit 1).
13. Subjects may be on intranasal steroid if it has been maintained for 4 weeks prior to screen and a constant stable dose is maintained for the duration of the trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To determine subject preference of a traditional paper symptom diary vs. the VOCEL® Mobile Diary. | 1 month

SECONDARY OUTCOMES:
Asthma symptom scores (Daytime/Nighttime), nocturnal awakenings, Peak expiratory flow rate (PEFR) and use of rescue medication (albuterol metered dose inhaler) as recorded by the subject on the traditional paper diary and the VOCEL® Mobile Diary. | 1 month
Change from baseline to end of treatment of peak expiratory flow. | 1 month
Change from baseline to end of treatment of FEV1. | 1 month
Determination of subject compliance with Alvesco® (ciclesonide), study medication dosing, as recorded on a traditional paper symptom diary and the VOCEL® Mobile Diary. | 1 month
Determination of patient generated assessment of ease of use of Alvesco® (ciclesonide) in regards to learning, daily use and difficulties experienced. | 1 month
Clinician generated assessment of the traditional paper diary and the VOCEL® Mobile Diary. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Eli O Meltzer, MD, Principal Investigator — Allergy & Asthma Medical Group & Research Center
Locations (1):
- Allergy & Asthma Medical Group & Research Center, San Diego, California, United States

REFERENCES:
- [Derived] Meltzer EO, Kelley N, Hovell MF. Randomized, cross-over evaluation of mobile phone vs paper diary in subjects with mild to moderate persistent asthma. Open Respir Med J. 2008;2:72-9. doi: 10.2174/1874306400802010072. Epub 2008 Sep 5. PMID 19412327